CLINICAL TRIAL: NCT03362684
Title: Ancillary Study of miR-31-3p and miR-31-5p Expression Levels in Patients Enrolled in the PETACC-8 Study, and of the Predictive Role of miR-31-3p Expression Level on Clinical Outcomes of Patients Treated With Cetuximab
Brief Title: PETACC-8 miR-31-3p and miR-31-5p Ancillary Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IntegraGen SA (Industry)
Collaborators: Federation Francophone de Cancerologie Digestive (Other); Exystat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IG2017001
Record Dates: First submitted 2017-11-24; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOX-4 plus Cetuximab (Experimental)
  Interventions: Drug: Cetuximab; Drug: FOLFOX
- FOLFOX-4 (Active Comparator)
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: Cetuximab — Cetuximab every 2 weeks
  Arms: FOLFOX-4 plus Cetuximab
Drug: FOLFOX — FOLFOX-4 every 2 weeks

SUMMARY:
This is a prospective-retrospective study to determine if the expression of the miRNA's miR-31-3p and miR-31-5p are prognostic of patient outcomes or predictive of the benefit from anti-EGFR therapy in stage III Colon Cancer. The present study will utilize FFPE tumor samples collected from patients enrolled in the PETACC-8 study conducted by the Fédération Francophone de Cancérologie Digestive (FFCD). This phase 3 clinical trial prospectively randomized fully resected stage III colon cancer patients to receive adjuvant treatment with either FOLFOX-4 plus cetuximab or FLOFOX-4 alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in PETACC08 study
* Signed informed consent for translational study
* FFPE tumor sample available for miR-31-3p and miR-31-5p expression testing

Exclusion Criteria:

* Patient who have withdrawn their consent for PETACC08 and/or for PETACC08 translational study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1808 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | From date of randomization until the date of first documented any signs or symptoms cancer relapse or date of death, whichever came first, assessed up to 7 years
  Difference in Disease Free Survival (DFS) for RAS/BRAF wild-type patients whose primary tumors have low miR-31-3p expression when treated with cetuximab plus FOLFOX-4 vs. FOLFOX-4 only .
Prognostic and predictive value of miR-31-3p expression on Disease Free Survival (DFS) | From date of randomization until the date of first documented any signs or symptoms cancer relapse or date of death, whichever came first, assessed up to 7 years
  If patients with RAS/BRAF wild-type (WT), low miR-31-3p expression tumors treated with cetuximab plus FOLFOX-4 arm have improved DFS vs. patients treated with FOLFOX-4 alone, the predictive and prognostic value of miR-31-3p expression level on cetuximab efficacy relative to DFS in patients with RAS/BRAF WT tumors .

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until date of death from any cause, assessed up to 7 years
  Difference in OS for RAS/BRAF wild-type patients whose primary tumors have low miR-31-3p expression when treated with cetuximab plus FOLFOX-4 vs. FOLFOX-4 only.
Prognostic and predictive value of miR-31-3p expression on OS | From date of randomization until date of death from any cause, assessed up to 7 years
  If patients with RAS/BRAF wild-type (WT), low miR-31-3p expression tumors treated with cetuximab plus FOLFOX-4 arm have improved OS vs. patients treated with FOLFOX-4 alone, the predictive and prognostic value of miR-31-3p expression level on cetuximab efficacy relative to OS in patients with RAS/BRAF WT tumors .
Survival after recurrence (SAR) | From date of the first documented recurrence to the date of death from any cause, assessed up to 7 years
  Difference in Survival after Recurrence (SAR) for RAS/BRAF wild-type patients whose primary tumors have low miR-31-3p expression when treated with cetuximab plus FOLFOX-4 vs. FOLFOX-4 only.
Prognostic and predictive value of miR-31-3p expression on SAR | From date of the first documented recurrence to the date of death from any cause, assessed up to 7 years
  If patients with RAS/BRAF wild-type (WT), low miR-31-3p expression tumors treated with cetuximab plus FOLFOX-4 arm have improved SAR vs. patients treated with FOLFOX-4 alone, the predictive and prognostic value of miR-31-3p expression level on cetuximab efficacy relative to SAR in patients with RAS/BRAF WT tumors .

OTHER OUTCOMES:
miR-31-3p cut-off | From the date of randomization until 7 years, or date of death from any cause.
  If pre-established cut-off for miR-31-3p expression does not achieve statistical significance, cut-off value of miR-31-3p expression that discriminates RAS Wild Type and BRAF Wild Type population treated with FOLFOX-4 + cetuximab in terms of DFS, OS and SAR.
miR-31-5p cut-off | From the date of randomization until 7 years, or date of death from any cause.
  Cut-off value for miR-31-5p expression which discriminates RAS Wild Type and BRAF Wild Type population treated with FOLFOX-4 + cetuximab in terms of DFS, OS and SAR.
Distribution of miR-31-5p expression | From the date of randomization until 7 years, or date of death from any cause.
  Distribution of miR-31-5p expression in the patient population and the correlation of miR-31-5p expression (quantitative) and of miR-31-5p expression level (low/high) with clinically significant co-variates and with the expression of miR-31-3p.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Taieb, MD, PhD, Principal Investigator — Hôpital Européen Georges-Pompidou; Pierre Laurent-Puig, MD, PhD, Principal Investigator — Hôpital Européen Georges-Pompidou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taieb J, Tabernero J, Mini E, Subtil F, Folprecht G, Van Laethem JL, Thaler J, Bridgewater J, Petersen LN, Blons H, Collette L, Van Cutsem E, Rougier P, Salazar R, Bedenne L, Emile JF, Laurent-Puig P, Lepage C; PETACC-8 Study Investigators. Oxaliplatin, fluorouracil, and leucovorin with or without cetuximab in patients with resected stage III colon cancer (PETACC-8): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Jul;15(8):862-73. doi: 10.1016/S1470-2045(14)70227-X. Epub 2014 Jun 11. PMID 24928083